CLINICAL TRIAL: NCT02529553
Title: A Phase 1 Study of LY3076226, a Fibroblast Growth Factor Receptor 3 (FGFR3) Antibody-Drug Conjugate, in Patients With Advanced or Metastatic Cancer
Brief Title: A Study of LY3076226 in Participants With Advanced or Metastatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15383; I7O-MC-JOBA (Other: Eli Lilly and Company)
Record Dates: First submitted 2015-08-19; First posted 2015-08-20 (Estimated); Results first posted 2020-04-17 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Advanced Cancer; Metastatic Cancer
Keywords: bladder cancer
MeSH Terms: conditions — Neoplasm Metastasis; Urinary Bladder Neoplasms | interventions — LY3076226

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LY3076226 (Experimental): Part A (dose escalation in advanced cancer): LY3076226 administered intravenously (IV) on day 1 of each 21 day cycle.
  Part B (dose expansion in advanced urothelial carcinoma): LY3076226 administered IV on day 1 of each 21 day cycle.
  Interventions: Drug: LY3076226

INTERVENTIONS:
Drug: LY3076226 — Administered IV

SUMMARY:
The main purpose of this study is to evaluate the safety of the study drug known as LY3076226 in participants with advanced or metastatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Have advanced or metastatic cancer and be an appropriate candidate for experimental therapy.

  * Part B: Have a diagnosis of bladder cancer.
  * Part B: Have alterations of FGFR3.
* Have adequate organ function.
* Have discontinued previous treatments for cancer and have resolution, except where otherwise stated in the inclusion criteria, of all clinically significant toxic effects of prior chemotherapy, surgery, or radiotherapy to Grade ≤1 by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), Version 4.0 (v 4.0).
* If participant is of reproductive potential, must agree to use medically approved contraceptive precautions during the study and for 3 months following the last dose of study drug. If the participant is a female of childbearing potential, must have had a negative serum or urine pregnancy test within 7 days of the first dose of study drug and must not be breastfeeding.

Exclusion Criteria:

* Have received treatment within 28 days of the initial dose of study drug with an investigational product or non-approved use of a drug or device (other than the study drug/device used in this study) or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study.
* Have preexisting corneal disease that may interfere with assessment for potential eye toxicity during the study.
* Have preexisting Grade ≥2 skin disorder (for example, erythema, dermatitis).
* Have serious preexisting medical conditions (left to the discretion of the investigator).
* Have symptomatic central nervous system (CNS) malignancy or metastasis (screening not required). Participants with treated CNS metastases are eligible for this study if they are not currently receiving corticosteroids and/or anticonvulsants, and their disease is asymptomatic and radiographically stable for at least 28 days.
* Have current acute or chronic leukemia.
* Have an active fungal, bacterial, and/or known viral infection including human immunodeficiency virus (HIV) or viral (A, B, or C) hepatitis (screening is not required).
* Have a second primary malignancy that, in the judgment of the investigator and sponsor, may affect the interpretation of results. Curatively treated nonmelanoma skin cancer or in situ carcinoma of any origin is allowed.
* Have Fridericia-corrected QT interval (QTcF) >480 milliseconds on screening electrocardiogram (ECG).
* Have a serious cardiac condition, such as congestive heart failure; New York Heart Association Class III/IV heart disease; unstable angina pectoris; myocardial infarction within the last 3 months; valvulopathy that is severe, moderate, or deemed clinically significant; or arrhythmias that are symptomatic or require treatment (not including participants with rate-controlled atrial fibrillation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-09; Primary Completion 2018-03-28 (Actual); Study Completion 2018-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (4):
- United States (3):
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - The START Center for Cancer Care, San Antonio, Texas
- For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Kollmannsberger C, Britten CD, Olszanski AJ, Walker JA, Zang W, Willard MD, Radtke DB, Farrington DL, Bell-McGuinn KM, Patnaik A. A phase 1 study of LY3076226, a fibroblast growth factor receptor 3 (FGFR3) antibody-drug conjugate, in patients with advanced or metastatic cancer. Invest New Drugs. 2021 Dec;39(6):1613-1623. doi: 10.1007/s10637-021-01146-x. Epub 2021 Jul 15. PMID 34264412
- See also: Click here for more information about this study: A Study of LY3076226 in Participants With Advanced or Metastatic Cancer — https://www.lillytrialguide.com/en-US/studies/solid-tumor/JOBA#?postal=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Part A (dose escalation in advanced cancer): LY3076226 administered intravenously (IV) on day 1 of each 21 day cycle.
  Part B (dose expansion in advanced urothelial carcinoma): LY3076226 administered IV on day 1 of each 21 day cycle.
Groups:
- LY3076226-0.2mg/kg: Part A cohort 1 of dose escalation of LY3076226 at 0.2 milligram per killogram (mg/kg).
- LY3076226-0.4mg/kg: Part A cohort 2 of dose escalation of LY3076226 at 0.4mg/kg.
- LY3076226-0.8mg/kg: Part A cohort 3 of dose escalation of LY3076226 at 0.8mg/kg.
- LY3076226-1.6mg/kg: Part A cohort 4 of dose escalation of LY3076226 at 1.6mg/kg.
- LY3076226-2.4mg/kg: Part A cohort 5 of dose escalation of LY3076226 at 2.4mg/kg.
- LY3076226-3.2mg/kg: Part A cohort 6 of dose escalation of LY3076226 at 3.2mg/kg.
- LY3076226-4.0mg/kg: Part A cohort 7 of dose escalation of LY3076226 at 4.0mg/kg.
- LY3076226-5.0mg/kg: Part A cohort 8 of dose escalation of LY3076226 at 5.0mg/kg.
- LY3076226-5.0mg/kg Dose Expansion: Part B dose expansion of LY3076226 at 5.0mg/kg.
Period: Overall Study
Arm/Group | LY3076226-0.2mg/kg | LY3076226-0.4mg/kg | LY3076226-0.8mg/kg | LY3076226-1.6mg/kg | LY3076226-2.4mg/kg | LY3076226-3.2mg/kg | LY3076226-4.0mg/kg | LY3076226-5.0mg/kg | LY3076226-5.0mg/kg Dose Expansion
Started | 1 | 1 | 1 | 3 | 3 | 4 | 3 | 6 | 3
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 1 | 1 | 3 | 3 | 4 | 3 | 6 | 3
Not completed — Progressive Disease | 1 | 0 | 1 | 3 | 2 | 3 | 3 | 5 | 3
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- LY3076226-0.2mg/kg: Part A cohort 1 of dose escalation of LY3076226 at 0.2mg/kg.
- Total: Total of all reporting groups
Arm/Group | LY3076226-0.2mg/kg | LY3076226-0.4mg/kg | LY3076226-0.8mg/kg | LY3076226-1.6mg/kg | LY3076226-2.4mg/kg | LY3076226-3.2mg/kg | LY3076226-4.0mg/kg | LY3076226-5.0mg/kg | LY3076226-5.0mg/kg Dose Expansion | Total
Number analyzed (Participants) | 1 | 1 | 1 | 3 | 3 | 4 | 3 | 6 | 3 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.0 | 73.0 | 56.0 | 68.3 (1.5) | 55.0 (6.2) | 63.0 (5.5) | 72.7 (9.8) | 65.8 (8.7) | 56.3 (5.9) | 63.0 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 2 | 2 | 4 | 2 | 2 | 1 | 13
  Male | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 4 | 2 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 6
  Not Hispanic or Latino | 0 | 1 | 1 | 2 | 2 | 3 | 2 | 5 | 3 | 19
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  White | 1 | 1 | 1 | 3 | 3 | 4 | 2 | 4 | 3 | 22
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 2 | 7
  United States | 1 | 1 | 1 | 3 | 1 | 3 | 2 | 5 | 1 | 18

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of LY3076226
Description: The MTD was defined as the highest dose tested that had less than 33% probability of causing a dose limiting toxicity (DLT).
Time Frame: Cycle 1 (21 Days)
Population: All participants enrolled in dose escalation.
Measure: Number; unit: milligrams
Groups:
- LY3076226: Part A dose escalation of LY3076226 administered intravenously (IV) on day 1 of cycle 1.
Arm/Group | LY3076226
Number analyzed (Participants) | 22
milligrams | 5.0

2. Secondary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY3076226
Time Frame: Predose: Day 1 (Cycle 1) and 63 (Cycle 3); Postdose: 0.05, 1, 3, 6, 24 and 72 hours
Population: All participants with adequate measurable PK concentrations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter(μg/mL)
Groups:
- LY3076226-0.2mg/kg: Cohort 1 of dose escalation of LY3076226 at 0.2 mg/kg.
- LY3076226-0.4mg/kg: Cohort 2 of dose escalation of LY3076226 at 0.4mg/kg.
- LY3076226-0.8mg/kg: Cohort 3 of dose escalation of LY3076226 at 0.8mg/kg.
- LY3076226-1.6mg/kg: Cohort 4 of dose escalation of LY3076226 at 1.6mg/kg.
- LY3076226-2.4mg/kg: Cohort 5 of dose escalation of LY3076226 at 2.4mg/kg.
- LY3076226-3.2mg/kg: Cohort 6 of dose escalation of LY3076226 at 3.2mg/kg.
- LY3076226-4.0mg/kg: Cohort 7 of dose escalation of LY3076226 at 4.0mg/kg.
- LY3076226-5.0mg/kg: Cohort 8 of dose escalation of LY3076226 at 5.0mg/kg.
- LY3076226-5.0mg/kg Dose Expansion: Dose expansion of LY3076226 at 5.0mg/kg.
Arm/Group | LY3076226-0.2mg/kg | LY3076226-0.4mg/kg | LY3076226-0.8mg/kg | LY3076226-1.6mg/kg | LY3076226-2.4mg/kg | LY3076226-3.2mg/kg | LY3076226-4.0mg/kg | LY3076226-5.0mg/kg | LY3076226-5.0mg/kg Dose Expansion
Number analyzed (Participants) | 1 | 1 | 1 | 3 | 3 | 4 | 3 | 6 | 3
Micrograms per milliliter(μg/mL)
  Cycle 1 | 5.35 | 10.6 | 23.3 | 41.9 (22.2) | 133 (123) | 77.4 (20.5) | 104 (9.37) | 119 (16.2) | 101 (22.3)
  Cycle 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 3 | 2 | 3 | 4 | 3
  Cycle 3 |  |  |  |  | 62.0 (34.0) | 89.8 (100) | 105 (8.26) | 144 (5.60) | 95.7 (22.1)

3. Secondary Outcome: PK: Area Under the Concentration-Time Curve (AUC) of LY3076226
Time Frame: Predose: Day 1 (Cycle 1) and 63 (Cycle 3); Postdose: 0.05, 1, 3, 6, 24 and 72 hours
Population: All participants with adequate measurable PK concentrations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg per day per mL(μg/day/mL)
Arm/Group | LY3076226-0.2mg/kg | LY3076226-0.4mg/kg | LY3076226-0.8mg/kg | LY3076226-1.6mg/kg | LY3076226-2.4mg/kg | LY3076226-3.2mg/kg | LY3076226-4.0mg/kg | LY3076226-5.0mg/kg | LY3076226-5.0mg/kg Dose Expansion
Number analyzed (Participants) | 1 | 1 | 1 | 3 | 3 | 4 | 3 | 6 | 3
μg per day per mL(μg/day/mL)
  Cycle 1 | 13.0 | 18.8 | 112 | 223 (14.3) | 503 (55.5) | 424 (33.2) | 665 (14.0) | 664 (29.5) | 638 (17.1)
  Cycle 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 3 | 2 | 3 | 4 | 3
  Cycle 3 |  |  |  |  | 374 (78.2) | 758 (833) | 688 (41.2) | 1120 (18.9) | 801 (27.0)

4. Secondary Outcome: Number of Participants With Tumor Response
Description: Tumor response was assessed using confirmed complete response (CR) or partial response (PR) according to Response Evaluation Criteria In Solid Tumors (RECIST version 1.1). Complete response (CR) was the disappearance of all target and non-target lesions and normalization of tumor marker levels of non-target lesions; partial response (PR) was at least a 30% decrease in the sum of the longest diameter of target lesions.
Time Frame: Baseline through Study Completion (Cycle 3, day 21)
Population: All enrolled participants.
Measure: Number; unit: participants
Arm/Group | LY3076226-0.2mg/kg | LY3076226-0.4mg/kg | LY3076226-0.8mg/kg | LY3076226-1.6mg/kg | LY3076226-2.4mg/kg | LY3076226-3.2mg/kg | LY3076226-4.0mg/kg | LY3076226-5.0mg/kg | LY3076226-5.0mg/kg Dose Expansion
Number analyzed (Participants) | 1 | 1 | 1 | 3 | 3 | 4 | 3 | 6 | 3
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up To 33 Days post study treatment
Description: All participants who received at least one dose of study drug.
Arm/Group | LY3076226-0.2mg/kg | LY3076226-0.4mg/kg | LY3076226-0.8mg/kg | LY3076226-1.6mg/kg | LY3076226-2.4mg/kg | LY3076226-3.2mg/kg | LY3076226-4.0mg/kg | LY3076226-5.0mg/kg | LY3076226-5.0mg/kg Dose Expansion
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1 | 0/1 | 0/3 | 0/3 | 0/4 | 0/3 | 0/6 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/1 | 1/1 | 0/1 | 1/3 | 1/3 | 0/4 | 0/3 | 1/6 | 0/3
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 1/1 | 3/3 | 3/3 | 4/4 | 3/3 | 6/6 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY3076226-0.2mg/kg (N=1) | LY3076226-0.4mg/kg (N=1) | LY3076226-0.8mg/kg (N=1) | LY3076226-1.6mg/kg (N=3) | LY3076226-2.4mg/kg (N=3) | LY3076226-3.2mg/kg (N=4) | LY3076226-4.0mg/kg (N=3) | LY3076226-5.0mg/kg (N=6) | LY3076226-5.0mg/kg Dose Expansion (N=3)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY3076226-0.2mg/kg (N=1) | LY3076226-0.4mg/kg (N=1) | LY3076226-0.8mg/kg (N=1) | LY3076226-1.6mg/kg (N=3) | LY3076226-2.4mg/kg (N=3) | LY3076226-3.2mg/kg (N=4) | LY3076226-4.0mg/kg (N=3) | LY3076226-5.0mg/kg (N=6) | LY3076226-5.0mg/kg Dose Expansion (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Corneal epithelial microcysts (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Keratitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Photopsia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Retinal pigment epitheliopathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 1 (1) | 3 (6) | 4 (4) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 3 (3) | 2 (2) | 0 (0) | 2 (2) | 2 (8)
Oesophageal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal discharge (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0)
Early satiety (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 3 (4) | 0 (0) | 2 (3)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Nasal vestibulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (3)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (2) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 2 (3) | 1 (2) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 1 (1)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chromaturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to pipeline reprioritization, development of LY3076226 was discontinued at the end of 2017 and no further patients were enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2015-08-06): https://cdn.clinicaltrials.gov/large-docs/53/NCT02529553/Prot_000.pdf
  • Statistical Analysis Plan (2015-06-24): https://cdn.clinicaltrials.gov/large-docs/53/NCT02529553/SAP_001.pdf